CLINICAL TRIAL: NCT04135131
Title: Comparison of The Efficacy of Pilates Exercises and Home Exercise Program on Pain, Functional Level and Thickness of Core Muscles in Patients With Low Back Pain
Brief Title: Efficacyof Pilates Exercises in Lowback Pain
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Duygu Geler Külcü, Clinical Professor, Head of Physical Therapy, Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HNEAH-KAEK 2017/kk/19
Record Dates: First submitted 2019-09-29; First posted 2019-10-22 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Low Back Pain; Physical Therapy; Pilates
Keywords: Abdominal Muscles; Exercise Therapy; Low back pain; Paraspinal Muscles
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Prospective, randomized-single blinded study
Masking Description: chronic low back pain patients, which has home exercises or pilates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PILATES MAT EXERCISE EFFECT ON LOW BACK PAIN (Experimental): Patients were randomized into pilates (group 1) or home exercise group (group 2) 3 times/week for 8 weeks. The evaluations were made at the beginning and end of the treatment. Outcome parameters were VAS, Oswestry Disability Index, Qubec Disability Scale, Short Form-36, Beck Depression Questionnaire, sit and reach, Modified Schöber and sit up tests. Multifidus and abdominal muscle thickness were measured by ultrasound image
  Interventions: Other: pilates mat exercises and home exercises
- HOME EXERCISE (Placebo Comparator): The exercise program included the pelvic tilt in the supine position, hamstring stretch, hip flexors and lumbar extensor stretch, bridge, strengthening the abdominal muscles, cat/camel exercises in the crawl position, leaning on the forearms in the prone position, strengthening the back extensors, and crossed-arms/legs lift exercises. Patients were asked to perform three sets of exercises (10 repetitions) for three times a week for 8 weeks. Exercise training was provided by a physiotherapist. Patients were also provided an illustrated exercise brochure along with an exercise diary to record the number of days on which exercise was performed. They were followed up by phone calls every 2 weeks
  Interventions: Other: pilates mat exercises and home exercises

INTERVENTIONS:
Other: pilates mat exercises and home exercises — Patients with low back pain were randomized into pilates (group 1) or home exercise group (group 2) 3 times/week for 8 weeks. Pilates mat exercise program comprised three sessions a week for 8 weeks (Monday, Wednesday, and Friday), with each session being scheduled for 1 h (5-min warm-up, 50-min exercise, and 5-min cooling) and each set comprising 10 repetitions. The home exercise program included the pelvic tilt in the supine position, hamstring stretch, hip flexors and lumbar extensor stretch, bridge, strengthening the abdominal muscles, cat/camel exercises in the crawl position, leaning on the forearms in the prone position, strengthening the back extensors, and crossed-arms/legs lift exercises.

SUMMARY:
OBJECTIVE: To investigate the effects of pilates exercise by training the muscles responsible for core stabilization in patients with chronic non-specific low back pain (CNLPB); considering pain, functional level, depression, quality of life, and muscle thickness measured by Ultrasound Imaging and to compare it with home based exercise.

MATERIAL AND METHODS: A prospective, randomized-single blinded study included 60 female patients with CNLBP aged 18-60 years. Patients were randomized into 2 groups. The first group (n=30) performed pilates 3 days/week for 8 weeks. Sessions lasted about one hour and supervised by a pilates trainer. The second group (n=30) was given home exercise program 3 times/week for 8 weeks, each session lasting one hour. The evaluations were made both at the beginning and end of the treatment. Evaluation parameters included VAS (visual analogue scale), Oswestry Disability Index, Qubec Disability Scale, Short Form-36 (SF-36), Beck Depression Questionnaire, sit and reach test, Modified Schöber test, sit up test. Multifidus and abdominal muscle thickness were measured by Ultrasonographic Imaging.

DETAILED DESCRIPTION:
A prospective, randomized-single blinded study included 60 female patients with CNLBP aged 18-60 years. Patients were randomized into 2 groups. The first group (n=30) performed pilates 3 days/week for 8 weeks. Sessions lasted about one hour and supervised by a pilates trainer. The second group (n=30) was given home exercise program 3 times/week for 8 weeks, each session lasting one hour. The evaluations were made both at the beginning and end of the treatment. Evaluation parameters included VAS (visual analogue scale), Oswestry Disability Index, Qubec Disability Scale, Short Form-36 (SF-36), Beck Depression Questionnaire, sit and reach test, Modified Schöber test, sit up test. Multifidus and abdominal muscle thickness were measured by Ultrasonographic Imaging.

ELIGIBILITY:
Inclusion Criteria:

* chronic non-specific low back pain for >3 months,
* visual analog scale (VAS) score of 3-6
* female patients aged 18-60 years,
* body mass index (BMI) within normal limits (18.5-24.9 kg/m²)
* ability to continue the program.

Exclusion Criteria:

* Malignancies,
* infections
* inflammatory diseases
* severe osteoporosis,
* arthritis
* metabolic bone diseases
* pregnancy
* cardiovascular diseases that limit effort capacity
* other musculoskeletal conditions that may impede attaining positions required in exercises
* a history of spinal surgery
* cognitive impairment.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
VISUAL ANALOGUE SCALE (VAS) for pain | 6 months
  pain (min-max:0-10) Higher scores correlate to higher intensity of pain
The Oswestry Disability Index | 6 months
  lowback functional disability The minimum score is 0% and the maximum score is 100%. Higher scores correlate to greater disability.
The Quebec Back Pain Disability Scale | 6 months
  low back pain The minimum score is 20 and the maximum score is 100. Higher scores correlate to greater disability.
Short Form-36 | 6 months
  (quality of life) questionnaire that covers eight health domains;Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Beck Depression Questionnaire | 6 months
  depression The minimum score is 0 and maximum score is 63. Higher scores indicate greater symptom severity.
Sit and reach test | 6 months
  flexibility
Modified Schöber and sit up tests | 6 months
  flexibility and endurance

CONTACTS AND LOCATIONS:
Locations (1):
- Haydarpaşa Numune Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No